CLINICAL TRIAL: NCT07260721
Title: Investigator-initiated Trial to Evaluate the Performance and Utility of a Single-lead Electrocardiogram Patch-based Telemetry System in Patients Requiring In-hospital Telemetry Electrocardiogram Monitoring During Hospitalization
Brief Title: Evaluation of a Single-lead ECG Patch-based Telemetry System for In-hospital Monitoring
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1-2025-0048
Record Dates: First submitted 2025-11-14; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Arrhythmias; Atrial Fibrillation; Ventricular Tachycardia; Supraventricular Tachycardia; Bradycardia; Telemetry; Patient Monitoring; Hospitalization
MeSH Terms: conditions — Arrhythmias, Cardiac; Atrial Fibrillation; Tachycardia, Ventricular; Tachycardia, Supraventricular; Bradycardia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MEMO-Cue (Experimental): Participants receive continuous in-hospital ECG monitoring using the MEMO-Cue system, which combines a single-lead patch device with real-time telemetry software. Monitoring lasts 12 hours to 8 days, and arrhythmia detection performance is compared with retrospective analysis using MEMO Care.
  Interventions: Device: MEMO-Cue-based telemetry monitoring

INTERVENTIONS:
Device: MEMO-Cue-based telemetry monitoring — In-hospital telemetry electrocardiogram monitoring using the MEMO-Cue system, which integrates a single-lead patch-type Holter device (MEMO Patch M) with a central monitoring software (MEMO-Cue) and an analysis platform (MEMO Care). Participants requiring continuous ECG telemetry during hospitalization are monitored for at least 12 hours and up to 8 days to evaluate the system's clinical utility and performance in real-time arrhythmia detection compared with retrospective analysis using MEMO Care.

SUMMARY:
"This investigator-initiated, prospective, single-center clinical study evaluates the performance and clinical utility of a single-lead electrocardiogram (ECG) patch-based telemetry system for hospitalized patients who require in-hospital telemetry ECG monitoring. The system integrates real-time centralized surveillance (MEMO-Cue) with post-hoc analytic review (MEMO-Care) using ECG signals recorded by the MEMO Patch M, aiming to enable timely recognition of clinically important arrhythmias and to inform treatment decisions under routine inpatient conditions.

Adults (≥19 years) indicated for continuous ECG monitoring during admission are enrolled after written informed consent, with a planned sample size of 100 to yield approximately 90 evaluable participants (10% anticipated dropout). The design does not include randomization or blinding. Study procedures include a screening visit (eligibility and baseline data), an inpatient monitoring period of at least 12 hours and up to 8 days with simultaneous MEMO-Cue monitoring and MEMO Patch M recording, and an end-of-visit assessment when MEMO-Care analytic results become available. Concomitant therapies deemed clinically necessary are permitted and documented, and adverse events are prospectively assessed.

Clinical utility endpoints quantify care impact and timeliness: (1) rate of treatment plan changes (e.g., initiation or modification of anticoagulants or antiarrhythmic drugs, cardioversion scheduling, device implantation, or other actions); (2) time to recognition (days) of major arrhythmias-atrial fibrillation (AF), ventricular tachycardia (VT), pause, ventricular premature complex (VPC), and supraventricular tachycardia (SVT)-based on MEMO-Cue alarms or MEMO-Care results with objective confirmation; (3) reduction ratio in recognition time when identified earlier by MEMO-Cue versus MEMO-Care; and (4) proportion of participants with shortened recognition time by MEMO-Cue.

Clinical performance endpoints assess detection characteristics and agreement between MEMO-Cue alarms and MEMO-Care findings: (1) clinical sensitivity (true positive / [true positive + false negative]); (2) precision, i.e., positive predictive value (true positive / [true positive + false positive]); and (3) positive concordance rate (proportion of MEMO-Care-detected arrhythmias alerted by MEMO-Cue). Safety is captured as treatment-emergent adverse events after device application, including device-related skin reactions, detachment, or signal dropouts, with severity graded per NCI-CTCAE v5.0 and relationship to device recorded.

By characterizing real-time patch-based telemetry alongside analytic review and its influence on diagnostic timing and management, the study aims to generate practical evidence supporting feasibility, reliability, and workflow compatibility of single-lead patch telemetry for in-hospital ECG monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 19 years or older who provide written informed consent for participation.
* Patients requiring in-hospital telemetry electrocardiogram monitoring during hospitalization.

Exclusion Criteria:

* Known hypersensitivity or allergic reaction to adhesives or hydrogel.
* Presence of skin wounds at the intended application site of the investigational device.
* Implanted cardiac electronic devices such as pacemakers, ICDs, or other CIEDs
* Current or past history of skin cancer, rash, dermatologic disorders, keloid formation, or skin injury.
* Any condition judged by the investigator to increase risk or make participation inappropriate.
* Cognitive impairment that precludes understanding of study information or voluntary consent.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Clinical decision change rate based on MEMO-Cue monitoring | From baseline (start of MEMO-Cue monitoring) to end of monitoring period, up to 8 days during hospitalization.
  Clinical utility will be evaluated by rate of change in treatment plans (%)
Clinical decision change rate based on MEMO-Cue monitoring | From baseline (start of MEMO-Cue monitoring) to end of monitoring period, up to 8 days during hospitalization.
  Clinical utility will be evaluated by time to recognition of major arrhythmias (days)
Clinical decision change rate based on MEMO-Cue monitoring | From baseline (start of MEMO-Cue monitoring) to end of monitoring period, up to 8 days during hospitalization.
  Clinical utility will be evaluated by reduction rate in arrhythmia recognition time (%)
Clinical decision change rate based on MEMO-Cue monitoring | From baseline (start of MEMO-Cue monitoring) to end of monitoring period, up to 8 days during hospitalization.
  Clinical utility will be evaluated by proportion of participants with shortened recognition time
Clinical decision change rate based on MEMO-Cue monitoring | From baseline (start of MEMO-Cue monitoring) to end of monitoring period, up to 8 days during hospitalization.
  Clinical performance will be assessed by clinical sensitivity (%)
Clinical decision change rate based on MEMO-Cue monitoring | From baseline (start of MEMO-Cue monitoring) to end of monitoring period, up to 8 days during hospitalization.
  Clinical performance will be assessed by precision (%)
Clinical decision change rate based on MEMO-Cue monitoring | From baseline (start of MEMO-Cue monitoring) to end of monitoring period, up to 8 days during hospitalization.
  Clinical performance will be assessed by positive concordance rate (%)

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No